CLINICAL TRIAL: NCT03506516
Title: Does Mixing Alcoholic Drinks Make Hangover Worse? A Randomized Controlled Trial in a Naturalistic Setting
Brief Title: Does Mixing Alcoholic Drinks Make Hangover Worse?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: VEK16028829
Record Dates: First submitted 2018-02-12; First posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Alcohol-Related Disorders
Keywords: alcohol, hangover
MeSH Terms: conditions — Alcohol-Related Disorders | interventions — Ethanol; Sarcoglycans

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single type (Experimental): Restricted to drinking only one type of alcohol
  Interventions: Dietary Supplement: Single type alcohol
- mixed type (Active Comparator): Drinking and mixing different types of alcohols freely
  Interventions: Dietary Supplement: Mixing alcohol

INTERVENTIONS:
Dietary Supplement: Mixing alcohol — Alcoholic beverages, different types
  Other Names: Ethanol
  Arms: mixed type
Dietary Supplement: Single type alcohol — Alcoholic beverages, different types
  Other Names: Ethanol
  Arms: single type

SUMMARY:
Does mixing alcohol make hangover worse?

DETAILED DESCRIPTION:
Hangover is the most commonly occurring morbidity associated with heavy drinking.

Our aim was to test the hypothesis that mixing alcoholic drinks as compared to drinking one type of alcohol only (beer, wine or spirits) associate with a higher alcohol intake and worse hangover.

ELIGIBILITY:
Inclusion Criteria:

* written and oral consent
* minimum 18 years old
* participating in Danish Health Research Retreat in Turkey 2016
* will consume alcoholic beverages

Exclusion Criteria:

* underage
* will not consume alcoholic beverages

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-05-20 (Actual); Primary Completion 2016-05-30 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Acute Hangover Severity Scale (AHSS) | Baseline
  AHSS is a 12-item alcohol hangover measurement tool recommended for application in hangover research with a predictive validity of 92.4 %, significantly higher than that of other hangover scales (Penning et al., 2012). Alcohol hangover was measured thrice the day after drinking; in the morning immediately after waking up, at midday, and in the afternoon. The individual participant assessed his or her own hangover the day after.

SECONDARY OUTCOMES:
Number of drinks | Baseline
  Total number of drinks defined as 12 g of alcohol consumed during evening
Acute Hangover Severity Scale (AHSS) 2 | after 4 hours
  AHSS is a 12-item alcohol hangover measurement tool recommended for application in hangover research with a predictive validity of 92.4 %, significantly higher than that of other hangover scales (Penning et al., 2012). Alcohol hangover was measured thrice the day after drinking; in the morning immediately after waking up, at midday, and in the afternoon. The individual participant assessed his or her own hangover the day after.
Acute Hangover Severity Scale (AHSS) 3 | after 8 hours
  AHSS is a 12-item alcohol hangover measurement tool recommended for application in hangover research with a predictive validity of 92.4 %, significantly higher than that of other hangover scales (Penning et al., 2012). Alcohol hangover was measured thrice the day after drinking; in the morning immediately after waking up, at midday, and in the afternoon. The individual participant assessed his or her own hangover the day after.

CONTACTS AND LOCATIONS:
Overall Officials: Ole G Christiansen, MD, Principal Investigator — Zealand University Hospital